CLINICAL TRIAL: NCT06343961
Title: To Evaluate the Value of Vitrectomy Combined With Sodium Fluorescein Angiography in the Diagnosis and Treatment of Vascular Retinal Diseases
Brief Title: Intraoperative Application of Fluorescein Sodium Angiography in Vascular Retinopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jie Zhong (Other)
Responsible Party: Sponsor-Investigator, Jie Zhong, Principal Investigator, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-76
Record Dates: First submitted 2024-03-11; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Vascular Retinopathy of Left Eye (Disorder); Vascular Retinopathy of Right Eye (Disorder); Diabetic Retinopathy; Retinal Vein Occlusion; Retinal Vasculitis; Vitreous Hemorrhage
Keywords: Intraoperative fluoroscopy; Fluorescein Angiography; laser; targeted retinal photocoagulation; retinal vascular disease
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Vein Occlusion; Retinal Vasculitis; Vitreous Hemorrhage

STUDY DESIGN:
Intervention Model Description: A total of 80 patients with vitreous hemorrhage diagnosed in Sichuan Provincial People's Hospital from January 2024 to December 2025 were selected. The number of included cases was calculated according to the minimum sample size of 200 patients with vitreous hemorrhage in our hospital, 95% confidence level and 5% confidence interval, and the calculated result was 79. The included cases were equally divided by random number method. 40 patients in the control group were given vitrectomy and other conventional operations such as retinal laser photocoagulation. In contrast group, 40 patients were given vitrectomy combined with intraoperative fluorescein angiography and other conventional operations such as retinal laser photocoagulation. The diagnosis rate of primary disease cause, observation rate of neovascularization and non-perfusion area, visual acuity, visual field, thickness of macular fovea and postoperative complications (ciliary detachment, secondary vitreous hemorrhage, neovascu
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- targeted retinal photocoagulation(TRP) (Experimental): TRP is a laser technology aimed at the peripheral non-perfusion and ischemic areas of the retina, and the laser area is determined according to the degree and progression ofthe patient's retinopathy.TRP can speciﬁcally act on unperfused retinal capillaries and retinal intermediate ischemic areas, reduce damage to tissue perfusion areas and panretinal photocoagulation (PRP) complications or adverse events.
  Interventions: Procedure: Intraoperative Fluorescein Angiography
- panretinal photocoagulation(PRP) (Experimental): The scope oftraditional PRP is mainly distributed in the middle and peripheral part of the retina, 1.5-2 optic disc diameters (DD) posteriorly from the optic disc and 2 DD temporally from the fovea,bounded by the superior and inferior vascular arches; forward to the ampulla of the vortex vein (or equator). Currently, PRP is the gold standard for the treatment of extensive areas of non-perfusion , as well as the main method for the treatment of severe nonproliferative diabetic retinopathy (NPDR) and PDR. However, due to the photochemical damage of the laser,panretinal laser photocoagulation causes more damage to the ocular tissue, and its side effects include hemorrhage, choroidal detachment, acute angle-closure glaucoma, etc. The occurrence of these complications is closely related to laser parameters such as increased duration and power and intensive treatment in a single session, which all lead to increased diffusion of thermal energy within the retina and choroid .
  Interventions: Procedure: Intraoperative Fluorescein Angiography

INTERVENTIONS:
Procedure: Intraoperative Fluorescein Angiography — Targeted laser photocoagulation under the guidance of intraoperative fluoroscopy

SUMMARY:
The study used a new surgical technique: intraoperative fluorescence imaging,In the 1980s, some scholars proposed the concept of intraoperative fluorescein angiography.During vitrectomy, intraoperative fluorescein angiography under 3D microscope can guide the surgeon to observe the non-perfusion area and new blood vessels on the same screen for accurate retinal photocoagulation therapy.Through this technology, the primary retinal disease can be identified in time after the removal of vitreous hemorrhage during surgery, providing effective imaging evidence support for the design of further treatment.

DETAILED DESCRIPTION:
With the improvement of living standards, the aging of population, the increasing incidence of chronic diseases such as hypertension and diabetes in China, the incidence of vascular retinopathy (retinal vein obstruction, diabetic retinopathy, retinal vasculitis, etc.) has also shown an increasing trend, and has become an important cause of blindness. Clinically, retinal angiofluciferin sodium angiography is mainly used to diagnose the cause of the disease. This technique has been widely used in clinic for more than 30 years, and it is safe and effective. However, its disadvantage is that patients need to have good refractive media, and the morphological changes of retinal blood vessels can be clearly observed. Vitreous hemorrhage is the most common complication of vascular retinal disease, which can be treated by vitrectomy. However, the occlusion of preoperative blood accumulation makes it impossible to effectively implement fluorescein sodium angiography, which makes doctors unable to make a comprehensive judgment of the disease in advance, which may affect the treatment plan and thus the therapeutic effect. Therefore, it is particularly important to comprehensively evaluate the primary disease of the patient's retina after removing the hematoma during the operation.

In the 1980s, some scholars proposed the concept of intraoperative fluorescein angiography, but due to poor camera resolution, insufficient digital image quality and transmission delay, the application of this technology in the surgical process is limited. In recent years, the rapid development of digitally assisted vitrectomy has enabled fundus surgeons to perform vitrectomy with a high-definition 3D screen. This technique also enables full visualization of intraoperative angiography that has not been possible before, and further real-time surgery based on this information. During vitrectomy, intraoperative fluorescein angiography under 3D microscope can guide the surgeon to observe the non-perfusion area and new blood vessels on the same screen for accurate retinal photocoagulation therapy. Through this technology, the primary retinal disease can be identified in time after the removal of vitreous hemorrhage during surgery, providing effective imaging evidence support for the design of further treatment. In this study, a specific light source and filter were designed according to Zeiss intraoperative microscope. Combined with 3D microscope, the morphology and function of retinal blood vessels can be effectively observed during the operation, which has not been reported in China. Using this technology, the team successfully observed clinical features such as non-perfusion area, neovascularization, and early formation of laser spots during vitrectomy, thus contributing to accurate treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* There is non-absorption vitreous hemorrhage in the target eye, which requires vitrectomy;
* can follow up according to the time specified by the study;
* Age ≥ 18 years old;
* Accurate Humphrey visual field test can be performed after surgery;
* Post-operative pupil dilation and clear media for laser photocoagulation, digital photography, and OCT scanning;

Exclusion Criteria:

* Active eyelid or accessory infection;
* Medical, surgical, panomental laser, or macular laser treatment of the study eye in the past 12 months;
* Brain disease, systemic immune system disease and other related medical history;
* Preoperative blood pressure (blood pressure greater than or equal to 180/110 mmHg), blood glucose (recent (past 6 months) or ongoing poor diabetes control, ·glycated hemoglobin > 10.0 mg/dl) poor control;
* Patients with choroidal detachment and ciliary detachment before surgery;
* Any systemic drug known to be toxic to the retina or associated with the risk of macular edema;Any prior eye conditions associated with the risk of macular edema;
* History of food and drug allergy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-18 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
best corrected visual acuity | 1 week, 1 month, 3 months, 6 months
  The best corrected visual acuity of patients at 1 week, 1 month, 3 months and 6 months after surgery
Central retinal thickness | 1 week, 1 month, 3 months, 6 months
  Central retinal thickness at 1 week, 1 month, 3 months, and 6 months after surgery